CLINICAL TRIAL: NCT04119726
Title: The Study Design of a Mobile Health (mHealth) Technology Associated Improvement of Drug Adherence in Patients With Acute Myocardial Infarction and Protocol for the Randomized, Controlled Trial（RESCIND-3)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Maoming People's Hospital (Other); Dongguan People's Hospital (Other Government); First People's Hospital, Shunde China (Other); Guangzhou Panyu Central Hospital (Other)
Responsible Party: Principal Investigator, Liu yong, Director, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: GDREC2018328H
Record Dates: First submitted 2019-10-07; First posted 2019-10-08 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Coronary Artery Disease
Keywords: Mobile health; Acute myocardial infarction; Cardioprotective medications; Randomized Controlled Trial
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: 400 patients with AMI on admission will be continuously enrolled and randomly allocated to either the control or intervention group. The intervention group will receive internet-based counseling, individual drug reminders, recommendations for healthy lifestyles, cardiovascular education about AMI, and follow-up reminders four times a week, while the control group will only receive cardiology knowledge and follow-up reminders four times a week. Mobile health tools (WeChat applet) were developed through cooperation with a technology company to establish appropriately. Trained research nurses will conduct the follow up in the 4th, 8th, 12th months by telephone or face-to-face visit. All the adverse events will be collected through a self-reported section in the mobile health tools. The study will evaluate the acceptability, utility of the intervention based on Internet consulting management.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research personnel, investigators, study coordinators and research assistants conducting the assessments and statisticians will not be informed of the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): The control group will receive a simplified tool including only the education message. The methodology will ensure that potential confounders by differences in nonspecific support and attention could be adjusted. Regular messages about prevention and cure of CHD will be sent to both groups four times a week. The short texts will be selected from the guidelines in China to avoid misinformation. There are also some pictures or videos that help patients change their behavior. Patients will be followed up for 4/8/12 months after admission through mHealth tools or telephone.
  Interventions: Behavioral: Usual Text Messages
- Intervention Group (Experimental): The intervention group will receive a complete social medial tool (web-based application ) installed on mobile phones including general education about coronary disease、personalized reminders and internet-based counseling. Patients will be followed up for 4/8/12 months after admission through mHealth tools or telephone.
  Interventions: Behavioral: Usual Text Messages; Behavioral: Personalized reminders; Behavioral: Internet-based counselling

INTERVENTIONS:
Behavioral: Usual Text Messages — Regular messages about prevention and cure of CHD will be sent to both groups four times a week. The short texts will be selected from the guidelines in China to avoid misinformation. There are also some pictures or videos that help patients change their behaviour.
Behavioral: Personalized reminders — Personal information, life behavior and risk factors will be registered when patients are enrolled. According to the baseline information, personalized knowledge will be sent to patients in the intervention group. Besides, patients will receive drug information and regular medication adherence reminders daily according to patients' baseline prescription drugs and modifications.
  Arms: Intervention Group
Behavioral: Internet-based counselling — The internet-based counselling is the key module of social media in the intervention group. The consultation content mainly includes the feedback of coronary heart disease secondary prevention drug compliance, the feedback of risk factor level control, the feedback of life and behaviour habits, the feedback of adverse events, the feedback of health education knowledge improvement, the reminders of data upload, behaviour change, and health education learning.
  When the patient has questions or discomfort during the medication, they can consult the applet and the applet will perform internet-based answers on the large database built by cardiologists. Meanwhile, social media will upload the question of consultation and report to the doctor according to individual differences in disease. If the patient is not satisfied with the auto-response, the patient can further consult his doctor and the doctor's response will be collected to improve the auto-response database
  Arms: Intervention Group

SUMMARY:
The RESCIND-3 study is a multicenter, double-blind, randomized controlled trial. It will be conducted in the departments of cardiology in 5 hospitals. Guangdong General Hospital ethics review board approved the study's design. 400 patients with AMI on admission will be continuously enrolled and randomly allocated to either the control or intervention group. The intervention group will receive internet-based counseling, individual drug reminders, recommendations for healthy lifestyles, cardiovascular education about AMI, and follow-up reminders four times a week, while the control group will only receive cardiology knowledge and follow-up reminders four times a week. Mobile health tools (WeChat applet) were developed through cooperation with a technology company to establish appropriate It will be blinding for investigators but all participants will be aware of whether their intervention is the 'experimental' treatment. Trained research nurses will conduct the follow up in the 4th, 8th, 12th months by telephone or face-to-face visit. All the adverse events will be collected through a self-reported section in the mobile health tools. The study will evaluate the acceptability, utility of the intervention based on Internet consulting management.

DETAILED DESCRIPTION:
Background：Antithrombotic drugs, β-blockers, statins and angiotensin converting enzyme inhibitor (ACEI)/angiotensin II receptor blockers (ARB) are recommended for patients with acute myocardial infarction(AMI). However, discontinuation of the drugs was associated with higher mortality. Few studies focused on the improvement of drug compliance through mHealth tools.

Objective：To investigate whether internet-based counseling could improve drug(Antithrombotic drugs, β-blockers, statins an ACEI/ARB) compliance following percutaneous coronary intervention(PCI) among patients with AMI within 1year's follow-up.

Study design：The study is a multicenter, randomized, prospective, double-blinded study. A total of 400 AMI patients following PCI will be randomized to intervention group or control group in addition to usual post-MI care. The intervention group will receive internet-based counseling, personalized reminders(drug information, healthy lifestyles advise) and educational message (cardiovascular knowledge and follow-up reminders) four times a week. It will be only usual messages (cardiovascular knowledge and follow-up reminders) supported four times a week in the control group. The primary endpoint is the discontinuation rate of coronary heart disease secondary prevention drugs (antiplatelet, ACEI/ARB, beta-blockers, and statins). The second endpoints include drug adherence scores assessed by the proportion of days covered(PDC) and major adverse cardiovascular events. Both groups will be followed up within 1year after PCI.

Summary：The multicentre randomized trial(RESCIND-3) will provide new evidence of the effectiveness of mHealth tools on improving 12-month drug compliance following PCI among patients with AMI.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Diagnosed with acute myocardial infarction
* Taking four kinds of cardioprotective medications(antiplatelet, ACEI/ARB, beta-blockers, and statins)
* Wechat and smartphone users
* Provide written informed consent

Exclusion Criteria:

* Pregnancy
* Malignant tumor or end-stage disease with a life expectancy of <1 year
* Unable to use mobile phone network applet
* Refuse to sign the informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Rate of discontinuation of drug | 1 year
  The discontinuation rate of each 4 kinds of coronary heart disease secondary prevention drug (antiplatelet drugs, ACEI/ARB, beta-blockers, and statins) without any professional permission. The continuous withdrawal time will be divided into three groups: ≤7 days, 8-30 days, more than 30 days.

SECONDARY OUTCOMES:
Acute myocardial infarction | 1 year
  Clinical evidence of acute myocardial injury(typical rise and fall of biochemical markers of myocardial necrosis to greater than twice the ULN or if markers were already elevated, further elevation of a marker to >50% of a previous value that was decreasing and >2× ULN, with ≥ 1 of the following) and myocardial ischemia, including: Myocardial ischemia; New ischemic ECG changes; Pathological Q wave appears; Imaging evidence and ischemic aetiology of new myocardium loss or abnormal local ventricular wall movement; Coronary thrombosis is determined by angiography or autopsy.
Medication discontinuance | 1 year
  Stop taking any one of antiplatelet drugs, β blockers, statins and ACEI/ARB without doctor's advice within one year of the onset of AMI.
Good drug compliance | 1 year
  It will be measured by the proportion of days covered (PDC) during one year following hospital discharge. Patients are classified as good compliance (PDC >80%) or no-good compliance (<80%) separately to each of the 4 preventive therapies.
Number of Participants with Major Adverse Cardiovascular Events. Target vascular revascularization (TVR) | 1 year
  All-cause mortality, defined as any death recorded between the date of the interview and the end of data linkage on 31 October 2016. Rehospitalization, stroke, target vascular revascularization (TVR). TVR is defined as any revascularization procedure (PCI or CABG) involving the vessel treated during the index PCI procedure for STEMI.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Liu, MD, Study Chair — Guangdong Cardiovascular Institute,Guangdong General Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China